CLINICAL TRIAL: NCT00174928
Title: A Phase 1, Single- and Repeated-Dose, Randomized, Open-Label, Multi-center Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Lansoprazole in Neonates With Clinically-Evident Gastroesophageal Reflux Disease.
Brief Title: A Study to Evaluate the Effect of Lansoprazole on Hospitalized Neonates With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP Clinical Sciences, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C03-042; U1111-1113-9957 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Pediatric GERD; Pediatric Gastroesophageal Reflux Disease; Neonates; lansoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole 0.5 mg/kg QD (Experimental)
  Interventions: Drug: Lansoprazole
- Lansoprazole 1.0 mg/kg QD (Experimental)
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 0.5 mg/kg/day suspension, orally, once daily for up to 5 days.
  Arms: Lansoprazole 0.5 mg/kg QD
Drug: Lansoprazole — Lansoprazole 1.0 mg/kg/day suspension, orally, once daily for up to 5 days.
  Arms: Lansoprazole 1.0 mg/kg QD

SUMMARY:
The purpose of this study is to understand how quickly lansoprazole, once daily (QD), improves feeding in premature babies or babies less than 28 days of age.

DETAILED DESCRIPTION:
A Phase 1, multi-center, pharmacokinetic/pharmacodynamic and safety, study in which neonates will be randomized in an open-label fashion to receive 5 days of open-label treatment with either lansoprazole pediatric suspension 1.0 mg/kg/day orally or lansoprazole pediatric suspension .5 mg/kg/day orally. On dosing Days 1 and 5, blood samples will be obtained for drug assay. All subjects will be evaluated for inclusion in the pH monitoring portion of the study and will undergo pH monitoring, provided it is clinically indicated, at the discretion of the investigator. Intragastric pH monitoring (up to 24 hours) will be performed at baseline, on dosing Day 1 (or Day 2) and on dosing Day 5 (or Day 6). Intraesophageal pH may be done in addition to intragastric pH at the discretion of the investigator. Subjects will be evaluated for safety, including a follow-up visit on post-dosing Day 14.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in the Neonatal Intensive Care or Special Care Nursery who have been fed orally or by feeding tube.
* Term or post-term infants with a body weight of >800 gms.
* Pre-term infants with a corrected age of less than 44 weeks.
* Clinically-evident GERD (feeding intolerance, regurgitation, wheezing or stridor with feedings)
* At least 7 days post-surgery without anticipated need for surgery during study
* No significant laboratory abnormalities

Exclusion Criteria:

* Unstable, clinically significant disease or abnormality
* Congenital anomaly of the upper gastrointestinal tract
* Clinical evidence of acute sepsis
* Cystic fibrosis
* Medical condition requiring subject to not be fed by mouth/gastric tube

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Analysis | Day 1 and 5
Mean Intragastric 24 hour pH (subset of six subjects) | Day -1, Day 1 and Day 5

SECONDARY OUTCOMES:
Gastroesophageal Reflux Disease Symptom Analysis | Days 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Result] Springer M, Atkinson S, North J, Raanan M. Safety and pharmacodynamics of lansoprazole in patients with gastroesophageal reflux disease aged <1 year. Paediatr Drugs. 2008;10(4):255-63. doi: 10.2165/00148581-200810040-00004. PMID 18590344
- [Result] Zhang W, Kukulka M, Witt G, Sutkowski-Markmann D, North J, Atkinson S. Age-dependent pharmacokinetics of lansoprazole in neonates and infants. Paediatr Drugs. 2008;10(4):265-74. doi: 10.2165/00148581-200810040-00005. PMID 18590345